CLINICAL TRIAL: NCT05475756
Title: Safety and Efficacy of Intrauterine Biological Barrier on Postoperative Adhesion After Hysteroscopic Adhesiolysis: a Prospective, Multicentre, Randomized, Positive Parallel Controlled, Non-inferiority, Clinical Trail
Brief Title: Safety and Efficacy of Intrauterine Biological Barrier on Postoperative Adhesion After Hysteroscopic Adhesiolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Zhangzhou Municipal Hospital of Fujian Province (Other); Guangzhou First People's Hospital (Other); Tang-Du Hospital (Other); Suzhou Municipal Hospital (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Limin Feng, Director of Obstetrics and Gynecology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RKM-GPSIS-CTP202201
Record Dates: First submitted 2022-06-07; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Intrauterine Adhesion
Keywords: Endometrium; Adhesion; Postoperative adhesion; Hysteroscopy; Biological Barrier; Adhesion prevention; Infertility; Hysteroscopic Adhesiolysis
MeSH Terms: conditions — Gynatresia; Tissue Adhesions; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Material：Small intestinal submucosa Specifications：A、B、C、D、E Dosage: investigator selects the specification and quantity(dosage) according to the postoperative uterine cavity volume Frequency：one time after the operation Duration：Single-use
  Interventions: Device: Intrauterine Biological Barrier
- Control Group (Active Comparator): Material: auto-crosslinked HA gel Specifications: 1 ml, 1.25 ml, 1.5 ml, 1.75 ml, 2 ml, 2.25 ml, 2.5 ml, 2.75 ml, 3 ml, 3.25 ml, 3.75 ml, 4 ml, 4.25 ml, 4.5 ml, 5 ml, 6 ml, 8ml Dosage: investigator selects the specification and quantity(dosage) according to the postoperative uterine cavity volume Frequency：one time after the operation Duration：Single-use
  Interventions: Device: Intrauterine Adhesion Barrier Gel

INTERVENTIONS:
Device: Intrauterine Biological Barrier — after Hysteroscopic adhesiolysis，use of Intrauterine Biological Barrier to repair uterine cavity
  Arms: Experimental Group
Device: Intrauterine Adhesion Barrier Gel — after Hysteroscopic adhesiolysis，use of Intrauterine Adhesion Barrier Gel to repair uterine cavity
  Arms: Control Group

SUMMARY:
To evaluate the safety and efficacy of Intrauterine Biological Barrier developed and produced by Chengdu TopRegMed Medical Technology Co., Ltd on postoperative adhesion after Hysteroscopic Adhesiolysis.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, parallel positive-control, non-inferior clinical trial, with the purpose to evaluate the efficacy and safety of Intrauterine Biological Barrier for the prevention or reduction of intrauterine adhesions after Hysteroscopic Adhesiolysis.

The trial will be conducted at six clinical centers with 264 subjects who meet all the inclusion/ exclusion criteria. Subjects will be randomly assigned to the experimental group and the control group in a 1:1 ratio. Subjects in the test group were treated with Intrauterine Biological Barrier (IBB) made by Chengdu TopRegMed Medical Technology Co. , Ltd. , while the patients in the positive control group were treated with commercially approved Intrauterine Adhesion Barrier Gel for uterine cavity made by Changzhou Bioregen biopharmaceutical Co. , Ltd. .

Subjects will be followed up for 12 months (360 days ± 30 days) after implantation. 73-days (± 12 days) after operation, the safety and effectiveness of IBB will be evaluated by demonstrating non-inferiority to commercially approved gel. If test group is non-inferiority, further study will be performed to explore whether the safety and effectiveness of the IBB is better than the control group in the aspect of the recurrence rate of intrauterine adhesion, types of intrauterine adhesion, postoperative endometrial repair, menstrual recovery and 1-year pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* （1）Age, yr20-40 (including boundary value), Female
* （2）Normal ovarian reserve function (FSH<10U/ml，AMH>2ng/ml)
* （3）Who suffered from moderate to severe intrauterine adhesions (AFS ≥ 5 points) diagnosed by hysteroscopy, and prepared to be treated by Hysteroscopic adhesiolysis
* （4）Both husband and wife have fertility intention during treatment
* （5）Accept to treatment and follow-up visits, Sign the ICF

Exclusion Criteria:

* （1）Severe systemic diseases, contraindications of surgical and cycle
* （2）Inflammation of reproductive tract, genital tuberculosis, pelvic infection, tumor of reproductive organs
* （3）Systemic diseases cause uterine bleeding
* （4）Allergic to hyaluronic acid or components
* （5）Allergic to swine sources medical device, or refuse to swine sources medical device for religious, ethnic and other reasons
* （6）Insufficient uterine cavity volume after Hysteroscopic adhesiolysis to place Intrauterine Biological Barrier or inject Intrauterine Adhesion Barrier Gel
* （7）Involved other clinical trial before Hysteroscopic adhesiolysis in 3 months or during the trail
* （8）Unable to tolerate anesthesia
* （9）Estrogen medicine was taken within 30 days of Hysteroscopic adhesiolysis
* （10）Other inadequacy patient assessed by the researchers

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-05-24 (Estimated); Study Completion 2025-05-23 (Estimated)

PRIMARY OUTCOMES:
Effective rate | Day 73±12
  At second-look hysteroscopy after Hysteroscopic adhesiolysis, the effective rate (%) = (number of cured + number of apparent effect)/total number in the group × 100%

SECONDARY OUTCOMES:
Recurrence rate of adhesions | Day 73±12
  The Presence of adhesions was determined at second-look hysteroscopy after Hysteroscopic adhesiolysis, and the recurrence rate of adhesions (%) = number of adhesion reoccurrence/total number in the group × 100%
Extent of uterine adhesions | Day 73±12
  The degree of uterine adhesions was assessed intraoperatively and at the second-look hysteroscopy with reference to the ESGE (European Society for Gynecological Endoscopy) criteria
Endometrial improvement | Day -7 to day 1, Day 100±10
  Endometrial thickness in millimeter and change values in millimeter by Ultrasonic Diagnostic Equipment Transvaginal Ultrasonic Probe Head at screening and visit 4
Time of menstrual recovery | Day 73±12
  Time to first menstruation after Hysteroscopic adhesiolysis
Duration of Menstrual recovery | Day 73±12, Day 100±10 , Day 180±30, Day 360±30
  Days of menstrual duration
Menstrual blood volume | Day 73±12, Day 100±10 , Day 180±30, Day 360±30
  Record and evaluate by Pictorial Blood Loss Assessment Chart (PBAC)
Pregnancy rate after operation 1year | Day 360±30
  Pregnancy rate (%) = number of pregnancies in the group/total number in the group × 100%

CONTACTS AND LOCATIONS:
Overall Officials: Limin Feng, Principal Investigator — Beijing Tiantan Hospital
Locations (6):
- China (6):
  - Anhui Provincial Hosptial, Hefei, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Guangzhou First people's Hospital, Guangzhou, Guangdong
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Tangdu Hospital, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No
No data sharing, only data collection and filling into paper CRF by each site

REFERENCES:
- [Background] March CM. Management of Asherman's syndrome. Reprod Biomed Online. 2011 Jul;23(1):63-76. doi: 10.1016/j.rbmo.2010.11.018. Epub 2010 Dec 4. PMID 21549641
- [Background] Yu D, Wong YM, Cheong Y, Xia E, Li TC. Asherman syndrome--one century later. Fertil Steril. 2008 Apr;89(4):759-79. doi: 10.1016/j.fertnstert.2008.02.096. PMID 18406834
- [Background] The American Fertility Society classifications of adnexal adhesions, distal tubal occlusion, tubal occlusion secondary to tubal ligation, tubal pregnancies, mullerian anomalies and intrauterine adhesions. Fertil Steril. 1988 Jun;49(6):944-55. doi: 10.1016/s0015-0282(16)59942-7. No abstract available. PMID 3371491
- [Background] Leone FP, Timmerman D, Bourne T, Valentin L, Epstein E, Goldstein SR, Marret H, Parsons AK, Gull B, Istre O, Sepulveda W, Ferrazzi E, Van den Bosch T. Terms, definitions and measurements to describe the sonographic features of the endometrium and intrauterine lesions: a consensus opinion from the International Endometrial Tumor Analysis (IETA) group. Ultrasound Obstet Gynecol. 2010 Jan;35(1):103-12. doi: 10.1002/uog.7487. PMID 20014360
- [Background] Higham JM, O'Brien PM, Shaw RW. Assessment of menstrual blood loss using a pictorial chart. Br J Obstet Gynaecol. 1990 Aug;97(8):734-9. doi: 10.1111/j.1471-0528.1990.tb16249.x. PMID 2400752
- [Background] AAGL Elevating Gynecologic Surgery. AAGL practice report: practice guidelines on intrauterine adhesions developed in collaboration with the European Society of Gynaecological Endoscopy (ESGE). Gynecol Surg. 2017;14(1):6. doi: 10.1186/s10397-017-1007-3. Epub 2017 May 1. No abstract available. PMID 28603474
- [Result] Kong D, Zhang L, Xu X, Zhang J, Li Y, Huang X. Small Intestine Submucosa Is a Potential Material for Intrauterine Adhesions Treatment in a Rat Model. Gynecol Obstet Invest. 2018;83(5):499-507. doi: 10.1159/000479086. Epub 2017 Jul 20. PMID 28723687
- [Result] Zhang X, Qiu J, Ding Y, Sun L, Hua K. Single port laparoscopy combined with vaginal cervicovaginal reconstruction in a patient with congenital atresia of the cervix. Fertil Steril. 2020 Mar;113(3):681-682. doi: 10.1016/j.fertnstert.2019.11.011. PMID 32192600
- [Result] Lin X, Wei M, Li TC, Huang Q, Huang D, Zhou F, Zhang S. A comparison of intrauterine balloon, intrauterine contraceptive device and hyaluronic acid gel in the prevention of adhesion reformation following hysteroscopic surgery for Asherman syndrome: a cohort study. Eur J Obstet Gynecol Reprod Biol. 2013 Oct;170(2):512-6. doi: 10.1016/j.ejogrb.2013.07.018. Epub 2013 Aug 7. PMID 23932377
- [Result] Amer MI, Abd-El-Maeboud KH, Abdelfatah I, Salama FA, Abdallah AS. Human amnion as a temporary biologic barrier after hysteroscopic lysis of severe intrauterine adhesions: pilot study. J Minim Invasive Gynecol. 2010 Sep-Oct;17(5):605-11. doi: 10.1016/j.jmig.2010.03.019. Epub 2010 Jun 23. PMID 20576472